CLINICAL TRIAL: NCT07127952
Title: Correlations of the Microvascular Abnormalities on NVC (Nail Fold Video Capillaroscopy) and GAVE (Gastric Antral Vascular Ectasia) as Seen on EGD
Acronym: GAVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Florentina Berianu, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-001900
Record Dates: First submitted 2025-07-29; First posted 2025-08-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Gastric Antral Vascular Ectasia
Keywords: GAVE; G.A.V.E; Gastric Antral Vascular; Gastric Antral Vascular Ectasia
MeSH Terms: conditions — Gastric Antral Vascular Ectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- GAVE with CTD (Other): Will include patients between 18 and 95 years old seen at Mayo Clinic in Florida who were diagnosed with GAVE (Gastric antral vascular ectasia) based on the EGD findings. Will include patients with gave and connective tissue disease. Patient can be identified using slicer dicer or advanced text explorer and will be invited to have a nail fold video capillaroscopy.
  Interventions: Device: Video Capillaroscopy
- GAVE without connective tissue disease (Other): Will include patients between 18 and 95 seen at Mayo Clinic in Florida who were diagnosed with GAVE based on the EGD findings. Will include patients with GAVE without connective tissue disease Patient can be identified using slicer dicer or advanced text explorer and will be invited to have a nail fold video capillaroscopy.
  Interventions: Device: Video Capillaroscopy

INTERVENTIONS:
Device: Video Capillaroscopy — A non-invasive imaging technique used to assess capillary structure and morphology in the nailfold area, commonly used in evaluating microvascular changes associated with connective tissue diseases.
  Other Names: Nailfold Video Capillaroscopy

SUMMARY:
The purpose of this research is to determine whether a procedure called capillaroscopy can help distinguish patients who are diagnosed with GAVE (gastric antral vascular ectasia) with an autoimmune disease versus idiopathic/other conditions based on EGD findings.

DETAILED DESCRIPTION:
The primary aim of this study is to define the prevalence and findings (as per quantification) of nail fold video capillaroscopy abnormalities in patients with GAVE. The secondary aim is to compare the findings of NVC and clinical presentation in patients with GAVE.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older with gave diagnosis as pair EGD performed in Gastroenterology as standard of care.

Patients with GAVE with connective tissue disease will be compared to patients with GAVE without a connective tissue disease.

Exclusion Criteria:

* Age less than 18 years of age, pregnant individuals, dialysis dependent, type 2 diabetes, recent hand trauma or manicure (<2 weeks), routine use of vibratory tools, history of acrocyanosis or erythromelalgia, previous diagnosis of a bleeding disorder, diagnosis of psoriasis, diagnosis of anti-phospholipid syndrome, exposure to toluene or benzoyl, diagnosis of psoriasis, diagnosis of COPD.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and Phenotypic with G.A.V.E | From enrollment to end of study once the accrual has been met within baseline of Day 1
  Defined the prevalence and phenotype of nail fold video capillaroscopy abnormalities in patients with G.A.V.E.

SECONDARY OUTCOMES:
Comparing Findings | From enrollment to end of study once the accrual has been met within baseline of day 1
  To compare the findings of and VC and clinical manifestation and organ involvement patients with gave and connective tissue disease to those with gave without connective tissue disease.

CONTACTS AND LOCATIONS:
Overall Officials: Florentina Berianu, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic (Florida), Jacksonville, Florida
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health Systems, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it has not been determined whether individual participant data (IPD) will be shared. The decision will depend on factors such as regulatory requirements, ethical considerations, and sponsor policies. If IPD sharing is implemented, appropriate safeguards will be in place to protect participant confidentiality.